CLINICAL TRIAL: NCT04144348
Title: A Phase 1b, Randomized, Observer-Blind, Placebo-Controlled, Dose Ranging Trial to Evaluate the Safety and Immunogenicity of mRNA-1653, a Combined Human Metapneumovirus (hMPV) and Parainfluenza Virus Type 3 (PIV3) Vaccine When Administered to Adults, and to Children 12 to 59 Months of Age With Serologic Evidence of Prior Exposure
Brief Title: Safety and Immunogenicity of mRNA-1653, a Combined Human Metapneumovirus (hMPV) and Parainfluenza Virus Type 3 (PIV3) Vaccine, in Healthy Adults, and Children 12 to 59 Months of Age With Serologic Evidence of Prior Exposure
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Prevention
Other Study IDs: mRNA-1653-P102
Record Dates: First submitted 2019-10-28; First posted 2019-10-30 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-01

CONDITIONS: Human Metapneumovirus and Human Parainfluenza Infection
Keywords: ModernaTX; mRNA-1653; human metapneumovirus; human parainfluenza; human parainfluenza vaccine; virus diseases; RNA virus infections; paramyxoviridae infections; mononegavirales infections
MeSH Terms: conditions — Virus Diseases; RNA Virus Infections; Paramyxoviridae Infections; Mononegavirales Infections | interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Parallel for the Adult Cohort, followed by Sequential Assignment for the Pediatric Cohort
Who Masked: Participant, Care Provider, Investigator
Masking Description: Observer blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- mRNA-1653, Adult participants (Experimental): Participants will receive 1 of 2 doses of mRNA-1653, administered via intramuscular injection, on Day 1 and Day 57.
  Interventions: Biological: mRNA-1653
- mRNA-1653 Pediatric participants (Experimental): Participants will receive 1 of 2 possible doses of mRNA-1653, administered via intramuscular injection, on Day 1 and Day 57.
  Interventions: Biological: mRNA-1653
- Placebo, Adult participants (Placebo Comparator): Participants will receive mRNA-1653-matching placebo, administered via intramuscular injection, on Day 1 and Day 57.
  Interventions: Biological: Placebo
- Placebo, Pediatric participants (Placebo Comparator): Participants will receive mRNA-1653-matching placebo, administered via intramuscular injection, on Day 1 and Day 57.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: mRNA-1653 — Sterile liquid for injection
  Arms: mRNA-1653 Pediatric participants; mRNA-1653, Adult participants
Biological: Placebo — Sterile liquid for injection
  Other Names: saline
  Arms: Placebo, Adult participants; Placebo, Pediatric participants

SUMMARY:
This clinical study will assess the safety and immunogenicity of 2 dose levels of mRNA-1653, a combined human metapneumovirus and human parainfluenza virus type 3 vaccine, in healthy adults (18 to 49 years of age) and 2 dose levels in children (12 to 59 months of age) with serologic evidence of prior exposure. The safety profile of the adult cohort will permit enrollment of the pediatric cohort.

ELIGIBILITY:
Key Inclusion Criteria:

* Adults 18 to 49 years of age and children 12 to 59 months of age at the time of consent who, in the opinion of the Investigator, are in good health based on review of medical history and screening physical examination
* Adult participant or parent(s)/legal guardian(s) has provided written informed consent for participation in this trial, including all evaluations and procedures as specified by this protocol
* Screening laboratory values Grade ≤1

Specific inclusion criteria for adults 18 to 49 years of age:

* Body mass index (BMI) from ≥18 kg/m^2 and ≤35 kg/m^2
* Female participants must be either of non-childbearing potential or if of childbearing potential may be enrolled if the participant: 1) has a negative pregnancy test at Screening and on the day of vaccination, and 2) has practiced adequate contraception or has abstained from all activities that could lead to pregnancy for 28 days prior to vaccination, and 3) has agreed to continue adequate contraception through 3 months following the last vaccination, and 4) is not currently breastfeeding

Specific inclusion criteria for children 12 to 59 months of age:

* Seropositive for both hMPV and PIV3 neutralizing antibody at Screening
* Has received routine immunizations appropriate for age per the Centers for Disease Control and Prevention (CDC) Advisory Committee on Immunization Practices (ACIP)
* Current height and weight above the third percentile for age

Key Exclusion Criteria:

Adult and pediatric participants eligible for this study must not meet any of the following criteria:

* Acutely ill or febrile (temperature ≥38.0℃/100.4°F, regardless of route) on the day of the first vaccination
* Any ongoing, symptomatic acute or chronic illness requiring medical or surgical care
* Receipt of, or plans for receipt of an inactivated vaccine(s) 14 days prior to though 14 days following each study injection or a live virus vaccine(s) within 28 days prior to, or plans to through 28 days following each study injection. The exception is any COVID-19 vaccine (regardless of type of vaccine) that becomes available to the participant during the study; efforts should be made to space study vaccinations and COVID-19 vaccinations by at least 7 and preferably 14 days, but COVID-19 vaccinations should not be delayed.
* Any chronic administration of an immunosuppressant or other immune modifying drug
* Prior administration of investigational agent using lipid nanoparticle formulations
* Donation of blood or blood products ≥450 mL within 28 days of the Screening visit (for the Adult Cohort)
* Intravenous blood products (red cells, platelets, immunoglobulins) within 3 months prior to enrollment
* Participated in an interventional clinical trial within 28 days prior to the day of enrollment, or plans to do so while enrolled in this trial
* Has a family member or household contact who is an employee of the research center or otherwise involved with the conduct of the study

Ages: 12 Months to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 51 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
Proportion of Participants with Solicited Local and Systemic Adverse Reactions (ARs) | Up to 7 days after each dose administration
Proportion of Participants with Unsolicited Adverse Events (AEs) | Up to 28 days after each dose administration
Proportion of Participants with Serious Adverse Events (SAEs) and Medically-Attended AEs | Up to 1 year after the last dose administration

SECONDARY OUTCOMES:
Geometric mean titer (GMT) of Serum Anti-hMPV and Anti-PIV3 Neutralizing Antibodies | Day 29, 57, 85, and 224 for adults; Day 29 and 85 for pediatric participants
Geometric Mean Ratio (GMR) of Post-Baseline/Baseline Titers of Serum Anti-hMPV and Anti-PIV3 Neutralizing Antibodies | Day 29, 57, 85, and 224 for adults; Day 29 and 85 for pediatric participants
Proportion of Participants with ≥2-Fold and ≥4-Fold Increases in Serum Anti-hMPV or Anti-PIV3 Neutralizing Antibody Titer from Baseline | Day 29, 57, 85, and 224 for adults; Day 29 and 85 for pediatric participants

CONTACTS AND LOCATIONS:
Locations (19):
- United States (19):
  - Central Research Associates Inc, Birmingham, Alabama
  - Meridian Clinical Research, Washington D.C., District of Columbia
  - Clinical Research Prime, Idaho Falls, Idaho
  - Heartland Research Associates LLC, El Dorado, Kansas
  - Heartland Research Associates LLC, Newton, Kansas
  - MedPharmics, Metairie, Louisiana
  - Meridian Clinical Research, LLC, Lincoln, Nebraska
  - Meridian Clinical Research, Norfolk, Nebraska
  - Meridian Clinical Research, LLC, Omaha, Nebraska
  - UHS Primary Care, Binghamton, New York
  - Child Healthcare Associates, Liverpool, New York
  - Child Healthcare Assoc., Syracuse, New York
  - Duke Vaccine and Trials Unit, Durham, North Carolina
  - Ohio Pediatric Research Assn Inc, Dayton, Ohio
  - Sanford Children's Hospital, Sioux Falls, South Dakota
  - Crossroads Clinical Research, Corpus Christi, Texas
  - University of Texas Medical Branch (UTMB), Galveston, Texas
  - Tekton Research Inc, San Antonio, Texas
  - Tanner Clinic, Layton, Utah

IPD SHARING:
Plan to Share IPD: No